CLINICAL TRIAL: NCT04037085
Title: Evaluation of PK/PD, Breastmilk Transfer, and Effectiveness of Ketamine After Cesarean Delivery - Part 1
Brief Title: Ketamine to Improve Recovery After Cesarean Delivery - Part 1
Acronym: KINETIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY18120046
Record Dates: First submitted 2019-02-02; First posted 2019-07-30 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Obstetric Pain; Postpartum Depression; Breastfeeding; Pain, Acute; Pain, Chronic; Obstetric Anesthesia Problems; Drug Effect; Opioid Use
MeSH Terms: conditions — Labor Pain; Depression, Postpartum; Breast Feeding; Acute Pain; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Prospective observational open-label trial (Part 1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): Ketamine - IV after cord clamping; IV infusion for 12 hours OR in the weaning population IV Ketamine infusion for 12 hours in the Montefiore CTRC
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Subjects in the intervention arm will receive infusion dosing as noted in arm/group descriptions at the time of cord clamping. Duration of infusion will be 12 hours. Concentrations of ketamine and ketamine metabolites (nor-ketamine, NKET; and dehydro-nor-ketamine, DHNK) are measured in maternal plasma and urine as well as breastmilk. Maternal side effects, adverse events, and efficacy endpoints will be measured over the 12 hour infusion and over 15 hours after infusion discontinuation.
  Other Names: Ketalar

SUMMARY:
The objective of this study is evaluate the breastmilk transfer and pharmacokinetics (Part 1) and effectiveness (Part 2) of a post-cesarean delivery intravenous ketamine bolus-and-infusion strategy, as a preventive analgesic modality to reduce pain and opioid requirements.

In Part 1, physiochemical analysis of pharmacokinetic/pharmacodynamic (PK/PD) and breastmilk transfer of ketamine and its metabolites will be assessed. Additionally calculated estimations for neonatal and infant exposure will be assessed.

In Part 2, PK/PD assessments will continue in a larger cohort; endpoints will also include postpartum pain, depression scores, central sensitization measures, patient-reported postpartum recovery scores, breastfeeding, and parent-infant bonding, assessed in the acute post-cesarean period and up to 12 weeks postpartum in a randomized controlled trial.

DETAILED DESCRIPTION:
Postpartum pain management strategies currently permit opioids for breakthrough pain, but strategies focused on minimizing or eliminating opioids are lacking. In the non-obstetric surgical population, modalities such as intravenous ketamine are well-recognized as effective adjuncts in opioid-reduction strategies for postoperative pain. Although there have been some studies of ketamine exposure in postpartum women without deleterious outcomes noted, these studies in pregnant and lactating women are limited by a lack of information on maternal pharmacokinetics, breastmilk secretion, and clinical effectiveness when used with standard multimodal analgesic approaches. There is also a lack of information on intermediate and long-term outcomes in this setting. This two-part trial will address these knowledge gap by advancing understanding of the safety and efficacy of ketamine and its metabolites in peripartum populations.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients (i.e., ≥18 years of age) and able to provide informed consent
* Cesarean Delivery, Scheduled or Non-Emergent (delivery within 15 minutes not necessary), or female weaning off of breastfeeding
* Cesarean cohort: ASA PS 2 or 3, with or without E designation (delivery within 15 minutes not necessary), Scheduled or Non-Emergent
* Spinal anesthesia with intrathecal morphine if Cesarean Delivery, Scheduled or Non-Emergent
* Multimodal postop analgesia with IV ketorolac, PO NSAID, and PO APAP if Cesarean Delivery, Scheduled or Non-Emergent
* Women who do not plan to breastfeed or who want to temporarily withhold breastfeeding or who are weaning off of breastfeeding (Part 1)

Exclusion Criteria:

* Cesarean Delivery under General Anesthesia
* Allergies to study medications
* ASA PS 4 or 4E
* ASA PS with E designation because delivery within 15 minutes required
* ASA PS greater than 4 (moribund patients)
* Contraindications to spinal anesthesia
* Contraindications to NSAIDs (gastric bypass, etc.)
* Contraindication to any other multimodal analgesia medicine
* Significant psychiatric history (depression and anxiety NOT exclusion criteria), uncontrolled hyperthyroidism, cardiac disease, fever, hypertension
* Adverse occurrence during caesarean section such as hemorrhage, need for transfusion, hemodynamic instability
* Placenta accreta spectrum or previa with large anticipated blood loss
* History of hallucinations, alcohol or illicit substance use/abuse, chronic opioid therapy, or chronic pain (chronic pain - defined by any condition requiring consistent follow up with pain specialist or daily administration of pain medications that could augment sedative effects)
* Pre-eclampsia with severe features

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Montefiore Hospital CTRC, Pittsburgh, Pennsylvania
  - Minhnoi C Wroble Biglan, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine: Ketamine - IV after cord clamping; IV infusion for 12 hours OR in the weaning population IV Ketamine infusion for 12 hours in the Montefiore CTRC
  Ketamine: Subjects in the intervention arm will receive bolus and infusion dosing as noted in arm/group descriptions at the time of cord clamping. Duration of infusion will be 12 hours. Breastmilk, maternal serum and urine, side effects, adverse events, and efficacy endpoints will be measured over the 12 hour infusion and over 15 hours after infusion discontinuation. For the weaning population, they will receive a 12 hour infusion in the CTRC and stay an additional 12 hours in the CTRC (or until discharged). Breastmilk, maternal serum and urine, side effects, adverse events, and efficacy endpoints will be measured over the 12 hour infusion and for 12 hours after infusion discontinuation.
Period: Overall Study
Arm/Group | Ketamine
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (3.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Number of pregnancies [Median (Full Range); unit: pregnancies] | 2 [1 to 5]
Parity [Median (Full Range); unit: live births] — Parity is the number of times a person has given birth to a live neonate.
  live births | 2 [1 to 5]
Maternal Weight [Mean (Full Range); unit: Kilograms (kg)] | 90.613 [53.8 to 137.4]

OUTCOME MEASURES:

1. Primary Outcome: Ketamine (AUC)
Description: Plasma will be used to calculate area under the plasma concentration-time curve (AUC 0-∞) of ketamine levels during infusion. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration of a dose of the drug.
Time Frame: 12 hour ketamine infusion
Measure: Mean (Standard Deviation); unit: mcg*min/mL
Arm/Group | Ketamine
Number analyzed (Participants) | 8
mcg*min/mL | 28.46 (9.97)

2. Primary Outcome: Steady State (Css)
Description: Ketamine steady state (Css) is defined as the concentration of drug in plasma at steady state.
Time Frame: 12 hours after ketamine infusion start
Measure: Number; unit: ng/mL
Arm/Group | Ketamine
Number analyzed (Participants) | 8
ng/mL | 35.58

3. Primary Outcome: Elimination Half Life (T1/2) for Ketamine
Description: Postpartum maternal plasma serum will be used to calculate postpartum maternal ketamine half-life (T1/2). b. Elimination half-life (t½) is the time required for drug concentration to decrease by one-half at the end drug dosing. Elimination half-life was obtained from the slope of terminal elimination phase.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Minutes | 364 (121)

4. Primary Outcome: Volume of Distribution Steady State (Vdss)
Description: Volume Distribution Steady State (Vdss) is the period of dynamic equilibrium of the drug calculated as the amount of drug in the body at time, t divided by the plasma concentration of the drug at time, t.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Liters | 1076 (617)

5. Primary Outcome: Ketamine Milk to Plasma Ratio (M:P)
Description: Milk to plasma ratio for KET were calculated by dividing the concentration of the respective components Ketamine in human milk by plasma concentration at the corresponding times (± 30 min). Ratios higher than 1 indicate breastmilk concentrations of ketamine and the metabolites would be higher in breastmilk than in maternal plasma concentrations.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Ratio | 3.15 (1.05)

6. Primary Outcome: Nor-ketamine Milk to Plasma Ratio
Description: Milk to plasma ratio of the Ketamine metabolite, Norketamine, calculated as the percentage of the maternal ketamine dose found from breastmilk. Milk to plasma ratio for NKET was calculated by dividing the concentration of the respective components Ketamine and Ketamine metabolites in human milk by plasma concentration at the corresponding times (± 30 min). Ratios higher than 1 indicate breastmilk concentrations of metabolites would be higher in breastmilk than in maternal plasma concentrations.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Ratio | 1.5 (0.19)

7. Primary Outcome: Hydroxynorketamine M:P Ratio
Description: Milk to plasma ratio of the Ketamine metabolite, Hydroxynorketamine, calculated as the percentage of the maternal ketamine dose found from breastmilk. Milk to plasma ratio for hydroxynorketamine was calculated by dividing the concentration of the respective ketamine metabolites in human milk by plasma concentration at the corresponding times (± 30 min). Ratios higher than 1 indicate breastmilk concentrations of the metabolites would be higher in breastmilk than in maternal plasma concentrations.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ketamine
Number analyzed (Participants) | 8
Ratio | 0.06 (0.015)

8. Primary Outcome: Relative Infant Dose of Ketamine (RID KET)
Description: Relative infant dose will be calculated as the percentage of the maternal ketamine dose found from breastmilk. The relative infant dose was calculated from the concentrations of ketamine in breast milk at different times following ketamine administration to the women. The concentration of ketamine was converted to amount by multiplying with the volume of breast milk collected at various time intervals. The cumulative dose of ketamine was calculated. An RID ≤10% was considered low.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: % Maternal ketamine in breastmilk
Arm/Group | Ketamine
Number analyzed (Participants) | 8
% Maternal ketamine in breastmilk | 0.0152 (0.02)

9. Primary Outcome: Relative Infant Dose of Ketamine Equivalent (Ketamine, Norketamine, Dehydro-norketamine)
Description: Relative infant dose (RID) will be calculated as the percentage of the maternal ketamine dose found from breastmilk. The relative infant dose was calculated from the concentrations of ketamine and its metabolites (ketamine, norketamine & dehydro-norketamine) in breast milk at different times following ketamine administration to the women.
Time Frame: 27 hours postpartum or 24 hour CTRC appointment for weaning population
Measure: Mean (Standard Deviation); unit: % maternal dose in breast milk
Groups:
- % RID Ketamine Equivalent (Ketamine, Norketamine, and Dehydronorketamine): Ketamine - IV after cord clamping; IV infusion for 12 hours OR in the weaning population IV Ketamine infusion for 12 hours in the Montefiore CTRC
  Ketamine: Subjects in the intervention arm will receive bolus and infusion dosing as noted in arm/group descriptions at the time of cord clamping. Duration of infusion will be 12 hours. Breastmilk, maternal serum and urine, side effects, adverse events, and efficacy endpoints will be measured over the 12 hour infusion and over 15 hours after infusion discontinuation. For the weaning population, they will receive a 12 hour infusion in the CTRC and stay an additional 12 hours in the CTRC (or until discharged). Breastmilk, maternal serum and urine, side effects, adverse events, and efficacy endpoints will be measured over the 12 hour infusion and for 12 hours after infusion discontinuation.
Arm/Group | % RID Ketamine Equivalent (Ketamine, Norketamine, and Dehydronorketamine)
Number analyzed (Participants) | 8
% maternal dose in breast milk | 0.0217 (0.027)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=8)
Light Headedness (Investigations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT04037085/Prot_003.pdf
  • Statistical Analysis Plan (2022-11-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT04037085/SAP_004.pdf
  • Informed Consent Form (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04037085/ICF_005.pdf